CLINICAL TRIAL: NCT05090046
Title: Understanding Neurocognitive Impairment After Trauma Exposure
Acronym: UNITE
Status: Completed | Type: Observational
Sponsor: University of Otago (Other)
Responsible Party: Sponsor
Other Study IDs: 11896201PQF
Record Dates: First submitted 2021-09-22; First posted 2021-10-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Trauma, Psychological; Earthquake
Keywords: Trauma; Earthquake; Cognitive impairment
MeSH Terms: conditions — Psychological Trauma; Wounds and Injuries; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be collected to assess the following biological markers:
  * Hormones (females only): progesterone, LH, FSH, testosterone, SHBG
  * Metabolic markers: total chol, HDL chol, LDL chol (calc), triglycerides, HbA1c
  * Inflammatory markers: CRP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Christchurch Health and Development Study (CHDS): The Christchurch Health and Development Study (CHDS) is a birth cohort study comprising 1265 people born in Christchurch in 1977. Participants have been followed to age 40, with 75-80% retention at data collection points.
  Interventions: Other: Trauma exposure

INTERVENTIONS:
Other: Trauma exposure — Exposure to the Canterbury earthquake sequence and other relevant psychological trauma

SUMMARY:
Individuals living in Canterbury (New Zealand) have experienced significant stress related to the Canterbury earthquake sequence. Previous research conducted at the Department of Psychological Medicine (Christchurch, New Zealand) has shown significant cognitive difficulties in a group of Cantabrians exposed to high levels of earthquake trauma. A high proportion (30%) perceive themselves to have significant cognitive difficulties, even seven years post-earthquake. People who perceive that they have cognitive difficulties find this distressing and tend to function less well in work and parenting. Understanding pathways underlying cognitive difficulties in the population is vital for developing appropriate treatments and strategies to help with this.

This will be the first study to investigate rates of, and factors contributing to, perceived cognitive difficulties in a large population exposed to multiple stressors and is important for the population of Canterbury, and populations affected by natural and man-made disasters worldwide.

Four hundred and sixty people who were exposed to the Canterbury earthquake sequence will be recruited from the Christchurch Health and Development Study (CHDS). Psychological, cognitive, functional and biological factors will be compared between those with the greatest levels of perceived cognitive difficulty and those with the lowest levels of difficulty. This will determine what factors relate most strongly to perceived cognitive difficulties, which will in turn be used to develop treatments for this population.

ELIGIBILITY:
Inclusion Criteria:

* Cohort member of the Christchurch Health and Development Study (born in 1977)
* Exposed to the Canterbury earthquake sequence
* In the highest or lowest quartile with regards to score on the Cognitive Failures Questionnaire

Exclusion Criteria:

* lifetime diagnosed psychotic disorder
* previous moderate to severe head injury (> 30 minutes loss of consciousness)
* current pregnancy
* intellectual disability (IQ < 80)
* residing outside of Canterbury

Ages: 44 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Christchurch Health and Development Study (CHDS) is a birth cohort study comprising 1265 people born in Christchurch in 1977. Participants have been followed to age 40, with 75-80% retention at data collection points. At the time of the February 2011 earthquake, 460 participants were in Christchurch and were subject to earthquake-related stresses.
  This study will recruit people from the CHDS who were exposed to the Canterbury earthquake sequence, based on results of an initial screening using the Cognitive Failures Questionnaire (CFQ): the quartile with the highest scores on the CFQ, and the quartile with the lowest scores will be selected and invited to attend a more comprehensive evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Subjective cognitive function | Past 6 months
  Assessed with the Cognitive Failures Questionnaire Minimum score = 0, maximum score = 100, higher scores reflect worse subjective cognitive function

SECONDARY OUTCOMES:
Global cognitive composite | Baseline
  Global cognitive composite will average Z-scores across the cognitive domains of (i) verbal learning and memory, (ii) visuospatial learning and memory, (iii) psychomotor speed, (iv) executive function, (v) working memory, (vi) sustained attention, and (vii) emotion processing. The Global cognitive composite score will be a single, averaged Z-value score, with a higher score reflecting better objective cognitive performance.
Verbal learning and memory | Baseline
  Z-scores from variables of the Rey Auditory Verbal Learning Test will be averaged to create a singe Z-score for the domain of 'Verbal Learning and Memory', with higher scores reflecting better performance.
Visuospatial learning and memory | Baseline
  Z-scores from variables of the Groton Maze Learning Test (CogState) will be averaged to create a singe Z-score for the domain of 'Visuospatial Learning and Memory', with higher scores reflecting better performance.
Psychomotor speed | Baseline
  Z-scores from variables of the Timed Chase Test (CogState), Trail Making Test - Part A, and Digit Symbol Coding Test will be averaged to create a singe Z-score for the domain of 'Psychomotor speed', with higher scores reflecting better performance.
Executive function | Baseline
  Z-scores from variables of the Trail Making Test - Part B and Category Fluency will be averaged to create a singe Z-score for the domain of 'Executive function', with higher scores reflecting better performance.
Working memory | Baseline
  Z-scores from variables of the Digit Span Test will be averaged to create a singe Z-score for the domain of 'Working memory', with higher scores reflecting better performance.
Sustained attention | Baseline
  Z-scores from variables of the Continuous Performance Test will be averaged to create a singe Z-score for the domain of 'Sustained attention', with higher scores reflecting better performance.
Facial emotion processing | Baseline
  Z-scores from variables of the Facial Expression Recognition Test and the Reading the Mind in the Eyes Test will be averaged to create a singe Z-score for the domain of 'Facial emotion processing', with higher scores reflecting better performance.
Rumination | Baseline
  Assessed with the Ruminative Responses Scale Minimum score = 25, maximum score = 100, higher scores reflect more severe rumination
Metacognitive beliefs | Baseline
  Assessed with the Metacognitions Questionnaire - 30-item version Minimum score = 30, maximum score = 120, higher scores reflect more problematic metacognitive beliefs Minimum score = 25, maximum score = 100, higher scores reflect more severe rumination
Psychosocial functioning | Past 2 weeks
  Assessed with the Social Adjustment Scale Minimum score = 1, maximum score = 5, higher scores reflect worse psychosocial functioning
Stressful life events | Past 5 years
  Number of stressful life events is assessed with the Life Events Scale (adapted from the Crisis in Family Systems - Revised Questionnaire) Minimum score = 0, higher score reflects more stressful life events
COVID-19 impact | Past 3 years
  Assessed with the COVID Psychosocial Impacts Scale (CPIS) Minimum score = 0, maximum score = 135, higher scores reflect more severe impact of COVID
Post-traumatic growth | Past 12 years
  Assessed with the Post-traumatic Growth Inventory (PTGI)
Mental health diagnoses | Baseline
  Assessed with the Mini International Neuropsychiatric Interview (MINI)
Metabolic markers | Baseline
  Blood levels of HbA1C, total cholesterol, HDL cholesterol, LDL cholesterol (calc), triglycerides
Inflammation | Baseline
  Blood levels of CRP
Sex hormones | Baseline
  Blood levels of progesterone, LH, FSH, testosterone, SHBG (females only)

OTHER OUTCOMES:
Data already obtained | 1977 to current
  Data will already be available from the CHDS database from birth to present, on the following relevant factors:
  * Childhood physical and emotional health
  * Childhood physical and sexual abuse
  * Previous stressful life event history
  * Lifetime mental health disorders
  * Traumatic brain injury
  * Environmental toxin exposure
  * Substance use
  * Personality factors (neuroticism, extraversion, novelty-seeking)
  * Educational achievement and IQ
  * Lifestyle factors, including diet and exercise
  * Parental functioning measures in childhood, including parental attachment and overprotection
  * Family functioning measures including parental maladaptive behaviour and illicit drug use, family instability, parental intimate partner violence
  * Trauma exposure in adulthood (including Christchurch earthquakes and Mosque shooting)
  * Menstrual history to identify those in early menopause The exact variables to be used for this study, and how they are to be aggregated, are TBC.

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Douglas, PhD, Principal Investigator — University of Otago
Locations (1):
- Department of Psychological Medicine, University of Otago, Christchurch, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Douglas K, Bell C, Tanveer S, Eggleston K, Porter R, Boden J. UNITE Project: understanding neurocognitive impairment after trauma exposure-study protocol of an observational study in Christchurch, New Zealand. BMJ Open. 2023 Aug 7;13(8):e072195. doi: 10.1136/bmjopen-2023-072195. PMID 37550025